CLINICAL TRIAL: NCT05035602
Title: Google Location History (GLH) as a Health Tool to Assess Physical Activity Profiles and Patterns Following Oesophagectomy and/or Gastrectomy
Brief Title: Google Location History Following Oesophagectomy and/or Gastrectomy
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 20SM6492
Record Dates: First submitted 2021-04-21; First posted 2021-09-05 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Oesophageal Cancer; Gastric Cancer; Survivorship; Quality of Life
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Oesophagectomy: Patients who have undergone oesophageal cancer resection.
  Interventions: Other: Physical activity assessment
- Gastrectomy: Patients who have undergone gastric cancer resection.
  Interventions: Other: Physical activity assessment
- Control group: A cohort consisting of healthy controls who have not been diagnosed with, or have undergone treatment for oesophageal or gastric cancer.
  Interventions: Other: Physical activity assessment

INTERVENTIONS:
Other: Physical activity assessment — Physical activity patterns will be obtained from google location history, using an Android phone

SUMMARY:
Surgery is the mainstay of treatment for patients with early-disease esophageal and gastric cancer. Open surgery for oesophageal cancer commonly involves large incisions in the chest, which is associated with a high rate of respiratory complications in the postoperative period. Patients with oesophageal or gastric cancer furthermore commonly present with significant weight loss, affecting both muscle mass and muscle strength. This could further decrease the physical fitness and increase the risk for experiencing complications after treatment. Patients also report a decreased physical functioning in quality of life at least 3 years after surgery, suggesting this is a persistent deficit. Currently, no long-term data is available assessing physical activity levels in oesophageal or gastric cancer survivors. Thus, quantifying physical activity levels in these patients may identify the period in which patients' activity levels are most likely to deteriorate. Activity levels will be assessed from Google Location History from the patient's phone, providing summary of physical activity over time. This information could be used in the future to provide adequate physical therapy intervention which might improve recovery in several aspects, such as physical fitness but also respiratory function and quality of life.

DETAILED DESCRIPTION:
Surgery is the mainstay of treatment for patients diagnosed with early-disease esophageal and gastric cancer. Open surgery for oesophageal cancer commonly involves large incisions in the chest, which is associated with a high rate of respiratory complications in the postoperative period. Several studies have shown that low physical activity levels are associated with increased risk for respiratory complication. Furthermore, patients with oesophageal or gastric cancer often present with significant weight loss, affecting both muscle mass and muscle strength. This could further decrease the physical fitness and increase the risk for experiencing complications after treatment. Moreover, open oesophagectomy involves thoracotomy, thus impairing respiratory mechanics with further deterioration in physical fitness. Patients also report a decreased physical functioning in quality of life at least 3 years after surgery, suggesting this is a persistent deficit. Currently, no long-term data is available assessing physical activity levels in oesophageal or gastric cancer survivors. Enhanced recovery programmes are evidence-based protocols aiming at early recovery after surgery with early mobilisation and physiotherapy, and have been shown to reduce respiratory complication rates. Thus, quantifying physical activity levels in these patients may identify the period in which patients' activity levels are most likely to deteriorate and whether these changes in physical activity are associated with changes in quality of life. Activity levels will be assessed from Google Location History from the patient's phone, providing summary of patterns of physical activity over time. This information could be used in the future to provide adequate physical therapy intervention which might improve recovery in several aspects, such as physical fitness but also respiratory function and quality of life.

ELIGIBILITY:
Inclusion Criteria post-oesophagectomy or -gastrectomy group:

* is 18 years or older, and below 90 years of age, AND
* be able to walk, run or cycle a short distance, AND
* has been diagnosed with or already treated for oesophageal or gastric cancer
* if already receiving treatment, any type of treatment is included, either surgical resection for early-stage disease or definitive chemotherapy for advanced disease, AND
* use and Android phone

Inclusion Criteria healthy controls:

* is 18 years or older, and below 90 years of age, AND
* no previous history of upper gastrointestinal cancer, AND
* not diagnosed with or undergoing treatment for active cancer since active cancer or cancer-related treatment might influence physical activity levels and quality of life, AND
* be able to walk, run or cycle a short distance, AND
* use an Android phone

Exclusion Criteria:

* lacks capacity or is unable to provide informed consent, OR
* below 18 years of age or over 90 years of age, OR
* cannot walk, run or cycle a short distance, OR
* is diagnosed with or undergoing treatment for active cancer other than oesophageal or gastric cancer, OR
* is pregnant, OR
* is not using an Android phone, as Google Location History data is only accessible from an Android device

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There will be three cohorts, consisting of post-oesophagectomy patients, post-gastrectomy patients and a third group consisting of healthy controls.
  The participants will be eligible if aged 18 years or older, up to 90 years of age.
  Participants will be eligible if they can provide informed consent and can walk, run or cycle a short distance, and if they are using an Android phone.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in physical activity pattern | Data will be collected up to 5 years prior to oesophageal or gastric cancer diagnosis and up to 5 years after oesophagectomy and/or gastrectomy.
  The physical activity pattern will be grouped into light vs moderate vigorous activity

SECONDARY OUTCOMES:
Presence of postoperative morbidity | Thirty-day postoperative morbidity will be collected.
  All types of postoperative morbidity will be assessed, including postoperative pulmonary complications, neurological damage, gastrointestinal symptoms, sepsis, anastomotic leak, cardiac or renal complications, urological complications, wound infection.
Health-related quality of life | Data will be collected at time of study recruitment, with HRQoL assessed at the time of recruitment (up to 5 years after surgery).
  The health-related quality of life will be reported using the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30.

OTHER OUTCOMES:
Self-reported physical activity | Data will be collected at time of study recruitment, up to 5 years after surgery.
  The self-reported physical activity will be estimated using the International Physical Activity Questionnaire (IPAQ)
Health-related Quality of Life | Data will be collected at time of study recruitment, up to 5 years after surgery.
  The Health-related Quality of Life will furthermore be reported using the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-OG25 questionnaire.
Health-related Quality of Life | Data will be collected at time of study recruitment, up to 5 years after surgery.
  The Health-related Quality of Life will furthermore be reported using the EuroQoL 5 dimensions, 5 level (EQ-5D-5L) questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All identifiable data will be anonymised. No data will be shared to other researchers outside the research team for the study.

REFERENCES:
- [Background] Costas-Chavarri A, Nandakumar G, Temin S, Lopes G, Cervantes A, Cruz Correa M, Engineer R, Hamashima C, Ho GF, Huitzil FD, Malekzadeh Moghani M, Sharara AI, Stern MC, Teh C, Vazquez Manjarrez SE, Verjee A, Yantiss R, Shah MA. Treatment of Patients With Early-Stage Colorectal Cancer: ASCO Resource-Stratified Guideline. J Glob Oncol. 2019 Feb;5:1-19. doi: 10.1200/JGO.18.00214. PMID 30802158
- [Background] Mariette C, Piessen G, Briez N, Gronnier C, Triboulet JP. Oesophagogastric junction adenocarcinoma: which therapeutic approach? Lancet Oncol. 2011 Mar;12(3):296-305. doi: 10.1016/S1470-2045(10)70125-X. Epub 2010 Nov 23. PMID 21109491
- [Background] Mariette C, Markar SR, Dabakuyo-Yonli TS, Meunier B, Pezet D, Collet D, D'Journo XB, Brigand C, Perniceni T, Carrere N, Mabrut JY, Msika S, Peschaud F, Prudhomme M, Bonnetain F, Piessen G; Federation de Recherche en Chirurgie (FRENCH) and French Eso-Gastric Tumors (FREGAT) Working Group. Hybrid Minimally Invasive Esophagectomy for Esophageal Cancer. N Engl J Med. 2019 Jan 10;380(2):152-162. doi: 10.1056/NEJMoa1805101. PMID 30625052
- [Background] Feeney C, Reynolds JV, Hussey J. Preoperative physical activity levels and postoperative pulmonary complications post-esophagectomy. Dis Esophagus. 2011 Sep;24(7):489-94. doi: 10.1111/j.1442-2050.2010.01171.x. Epub 2011 Feb 10. PMID 21309920
- [Background] Toriumi T, Yamashita H, Kawasaki K, Okumura Y, Wakamatsu K, Yagi K, Aikou S, Nomura S, Seto Y. Preoperative Exercise Habits are Associated with Post-gastrectomy Complications. World J Surg. 2020 Aug;44(8):2736-2742. doi: 10.1007/s00268-020-05493-3. PMID 32306081
- [Background] Wang L, Wang C, Guan S, Cheng Y. Impacts of physically active and under-active on clinical outcomes of esophageal cancer patients undergoing esophagectomy. Am J Cancer Res. 2016 Jul 1;6(7):1572-81. eCollection 2016. PMID 27508099
- [Background] Anandavadivelan P, Lagergren P. Cachexia in patients with oesophageal cancer. Nat Rev Clin Oncol. 2016 Mar;13(3):185-98. doi: 10.1038/nrclinonc.2015.200. Epub 2015 Nov 17. PMID 26573424
- [Background] Fukuda Y, Yamamoto K, Hirao M, Nishikawa K, Maeda S, Haraguchi N, Miyake M, Hama N, Miyamoto A, Ikeda M, Nakamori S, Sekimoto M, Fujitani K, Tsujinaka T. Prevalence of Malnutrition Among Gastric Cancer Patients Undergoing Gastrectomy and Optimal Preoperative Nutritional Support for Preventing Surgical Site Infections. Ann Surg Oncol. 2015 Dec;22 Suppl 3:S778-85. doi: 10.1245/s10434-015-4820-9. Epub 2015 Aug 19. PMID 26286199
- [Background] Stewart GD, Skipworth RJ, Fearon KC. Cancer cachexia and fatigue. Clin Med (Lond). 2006 Mar-Apr;6(2):140-3. doi: 10.7861/clinmedicine.6-2-140. No abstract available. PMID 16688969
- [Background] Guinan EM, Bennett AE, Doyle SL, O'Neill L, Gannon J, Foley G, Elliott JA, O'Sullivan J, Reynolds JV, Hussey J. Measuring the impact of oesophagectomy on physical functioning and physical activity participation: a prospective study. BMC Cancer. 2019 Jul 12;19(1):682. doi: 10.1186/s12885-019-5888-6. PMID 31299920
- [Background] Lagergren P, Avery KN, Hughes R, Barham CP, Alderson D, Falk SJ, Blazeby JM. Health-related quality of life among patients cured by surgery for esophageal cancer. Cancer. 2007 Aug 1;110(3):686-93. doi: 10.1002/cncr.22833. PMID 17582628
- [Background] Markar SR, Karthikesalingam A, Low DE. Enhanced recovery pathways lead to an improvement in postoperative outcomes following esophagectomy: systematic review and pooled analysis. Dis Esophagus. 2015 Jul;28(5):468-75. doi: 10.1111/dote.12214. Epub 2014 Apr 3. PMID 24697876